CLINICAL TRIAL: NCT02439203
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Crossover Study in Subjects With Parkinson's Disease With Moderate to Severe Levodopa-induced Dyskinesia, to Assess the Efficacy, Safety/Tolerability and Pharmacokinetics of JM-010
Brief Title: Efficacy and Safety of JM-010 in PD With Levodopa-Induced Dyskinesia
Acronym: LID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Collaborators: Contera Pharma ApS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JM-010CS01
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease; Levodopa Induced Dyskinesia (LID)
Keywords: Parkinson Disease; Levodopa Induced Dyskinesia (LID); Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JM-010 (Experimental): JM-010
  Interventions: Drug: JM-010
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JM-010
  Arms: JM-010
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of a randomized, double-blind, placebo-controlled, 2-way crossover study is to evaluate the efficacy, safety/tolerability and pharmacokinetics of JM-010 for the treatment of subjects with Parkinson's Disease (PD) with levodopa-induced dyskinesia (LID).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Subject with a diagnosis of moderate to severe idiopathic PD with showing responsiveness to levodopa.
* All anti-Parkinsonian medications and levodopa must be stable for at least 1 week prior to the start of the run-in period.
* Subject with stable predictable peak-effect LID of at least 2 hours of the awake day and with at least moderately disabling.
* Amantadine and/or monoamine oxidase (MAO) inhibitor must be stopped at least 2 weeks prior to the start of Treatment Period 1(TP 1).

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other Parkinsonian syndromes exists, such as secondary Parkinsonism, Parkinson-plus syndromes or other neurological degenerative diseases.
* History of any other brain surgery or surgery for the treatment of PD.
* Current primary psychiatric diagnosis of acute psychotic disorder or other primary psychiatric diagnoses.
* A history of psychosis and/or treatment with antipsychotics within 3 months prior to the start of Treatment Period 1(TP1).
* A history of, or current, seizure disorders and subjects requiring treatment with anti-convulsants.
* Clinically significant abnormal laboratory data at screening.
* Clinically relevant ischemic heart symptoms or history of myocardial infarction, coronary artery bypass surgery or percutaneous transluminal coronary angioplasty, within the previous 12 months prior to the start of TP1.
* History of cerebrovascular accident or transient ischemic attack, coronary vasospasm/Prinzmetal's angina.
* History of serotonin syndrome.
* Breast feeding or pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Investigator-rated change in dyskinesia severity as assessed by the Abnormal Involuntary Movement Scale (AIMS) | 7 Days
  Investigator-rated change in dyskinesia severity as assessed by the AIMS after levodopa challenge

SECONDARY OUTCOMES:
Investigator-rated Parkinsonian disability using Unified Parkinson's Disease Rating Scale (UPDRS) Part III | 7 Days
  Investigator-rated Parkinsonian disability using UPDRS Part III after levodopa challenge
Subject-rated change in PD effects as assessed through daily Dyskinesia Questionnaires | Daily
  Subject-rated change in PD effects as assessed through daily dyskinesia questionnaires
Subject-rated change in dyskinesia severity as assessed by the Clinical Global Impression (CGI) scale | 7 Days
  Subject-rated change in dyskinesia severity as assessed by the CGI scale
Safety and Tolerability as measured by assessment of abnormalities in physical examinations, safety laboratory examinations, 12-lead electrocardiogram (ECG) and vital signs; collection of adverse events (AEs) | 28 Days
  Assessment of abnormalities in physical examinations, safety laboratory examinations, 12-lead electrocardiogram (ECG) and vital signs; collection of adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Bloemfontein, South Africa